CLINICAL TRIAL: NCT02872350
Title: Prognostic Contribution of Abdominal Ultrasound in Necrotizing Enterocolitis in Preterm Infants Less Than 33SA.
Acronym: ECUN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-34; 2015-A01628-41 (Registry Identifier: IDRCB)
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: the Necrotizing Enterocolitis; Preterm Infants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Premature with necrotizing enterocolitis (Experimental)
  Interventions: Device: Abdominal ultrasound

INTERVENTIONS:
Device: Abdominal ultrasound — Techniques and predictive characteristics of the combination abdominal ultrasound abdomen and shot in the prognostic assessment of ECUN in premature under 33SA.

SUMMARY:
Enterocolitis necrotizing (ECUN) is a common and serious gastrointestinal disease in premature infants.

The diagnosis of ECUN based on clinical and radiological criteria. The abdomen plain film to date is the reference examination to confirm or refute the diagnosis. Indeed, the presence of pathognomonic signs (pneumatosis, aéroportie) on the abdomen of cliché can confirm the diagnosis. The prognostic value of these radiographic findings is currently controversial.

Abdominal ultrasound is a test whose possibilities in diagnostic and prognostic term began to be considered for some years. It also has other advantages, including that of not being a radiating examination. Studies on the prognostic value of abdominal ultrasound are rather few. Moreover, they involve a series of heterogeneous patients in terms of gestational age. Or the pathophysiology of ECUN in children born at term and in children born prematurely is not the same.

The objective is to study prospectively the prognostic contribution of abdominal ultrasound in the ECUN in premature under 33SA.

ELIGIBILITY:
Inclusion Criteria:

* Birth Term strictly less than 33SA
* Gestational age some (assessed on early ultrasound dating)
* Congenital malformation of Absence
* Suggestive clinical symptomatology of ECUN defined by the presence of abdominal bloating, increased residues (> 20% of the volume of enteral feeding) and the presence of blood in stool (macro- or microscopic)
* Radiologic investigation with a radiograph of abdomen and abdominal ultrasound done for the episode of ECUN
* Maximum interval between imaging tests 2 hours
* No parental opposition to the participation of children in the study

Exclusion Criteria:

* Term higher or equal to 33 weeks
* Congenital malformation
* Parental Opposition (or legal representatives) to participate in the study

Max Age: 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 95 (Estimated)
Dates: Start 2016-10; Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Comment prognostic evaluation by abdominal ultrasound | 36 months
  Assessment in clinical outcome prognosis by abdominal ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No